CLINICAL TRIAL: NCT05582564
Title: The Effect of Newspaper Reporting on COVID-19 Vaccine Hesitancy: a Randomised Controlled Trial
Acronym: COVANEW
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bari Aldo Moro (Other)
Responsible Party: Principal Investigator, Anna Rinaldi, Assistant Professor, University of Bari Aldo Moro
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 00001
Record Dates: First submitted 2022-10-13; First posted 2022-10-17 (Actual); Last update posted 2022-10-17 (Actual); Status verified 2022-10

CONDITIONS: Vaccine Hesitancy
Keywords: vaccine hesitancy
MeSH Terms: conditions — Vaccination Hesitancy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- concrete text (Other): Italian and French unvaccinated cohorts (n= 164; n=163)
  Interventions: Other: abstract vs concrete texts
- abstract text (Other): Italian and French unvaccinated cohorts (n=155; n=153)
  Interventions: Other: abstract vs concrete texts
- abstract task (Other): Italian and French unvaccinated cohorts (n=54; n=55)
  Interventions: Other: abstract vs concrete texts
- concrete task (Other): Italian and French unvaccinated cohorts (n=55; n=56)
  Interventions: Other: abstract vs concrete texts
- control (Other): Italian and French unvaccinated cohorts (n=103; n=110)
  Interventions: Other: abstract vs concrete texts

INTERVENTIONS:
Other: abstract vs concrete texts — The main experiment involved two groups of participants and two different articles about vaccine-related thrombosis taken from two Italian newspapers. One article used a more abstract descriptive style and language, while the other used a more anecdotical style and concrete language: each group read only one of these articles. Both articles are the same length and describe an episode of vaccine-related thrombosis. The abstract text uses a more formal and impersonal language, reporting more scientific considerations; the concrete text uses a more familiar and emotional style and provides a more anecdotical description of the case. Texts were also weighted according to a concreteness semantic vocabulary. French received translated versions.Two other groups were assigned categorization tasks; one was asked to complete a concrete categorization task and the other an abstract categorization task.
  Other Names: abstract vs concrete tasks

SUMMARY:
COVID-19 vaccine hesitancy can be observed at different rates in different countries. 1,068 people were surveyed in France and Italy to inquire about individual potential acceptance, focusing on time preferences, in a risk-return framework: having the vaccination today, in a month, and in 3 months; perceived risks of vaccination and COVID-19; and expected benefit of the vaccine. A randomized controlled trial was conducted to understand how everyday stimuli, such as fact-based news about vaccines, impact on audience acceptance of vaccination. The main experiment involved two groups of participants and two different articles about vaccine-related thrombosis taken from two Italian newspapers. One article used a more abstract description and language, and the other used a more anecdotical description and concrete language; each group read only one of these articles. Two other groups were assigned categorization tasks; one was asked to complete a concrete categorization task and the other an abstract categorization task.

DETAILED DESCRIPTION:
The goal of this RCT is to learn how journalistic news can affect vaccine hesitancy. 2 cohorts of unvaccinated individual, one Italian, one French. 5 arms design:

1. participants reading a fact-based newspaper article written in an abstract language
2. participants reading a fact-based newspaper article written in a more concrete language
3. participants performing abstract categorization task
4. participants performing concrete categorization task
5. control group answering questionnaire

Research questions:

i) Does a more abstract vs concrete language increase the willingness to receive the vaccine? ii) Does a more abstract vs concrete mindset increase the willingness to receive the vaccine? iii) Is a gender effect detectable?

ELIGIBILITY:
Inclusion Criteria:

unvaccinated individuals

Exclusion Criteria:

vaccinated individuals

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1068 (Actual)
Dates: Start 2021-06-02 (Actual); Primary Completion 2021-06-20 (Actual); Study Completion 2022-01-31 (Actual)

PRIMARY OUTCOMES:
vaccine hesitancy; number of participants accepting the vaccination | same day
  revealed preferences

CONTACTS AND LOCATIONS:
Locations (1):
- University of Bari Aldo Moro, Bari, Italy

IPD SHARING:
Plan to Share IPD: No
No personal data have been collected. Individual responses to the questionnaire will be shared without personal information of respondents on a public repository.

REFERENCES:
- [Background] Liberman N, Trope Y. Traversing psychological distance. Trends Cogn Sci. 2014 Jul;18(7):364-9. doi: 10.1016/j.tics.2014.03.001. Epub 2014 Apr 10. PMID 24726527
- [Background] Trope Y, Liberman N. Temporal construal. Psychol Rev. 2003 Jul;110(3):403-21. doi: 10.1037/0033-295x.110.3.403. PMID 12885109
- [Background] Loomba S, de Figueiredo A, Piatek SJ, de Graaf K, Larson HJ. Measuring the impact of COVID-19 vaccine misinformation on vaccination intent in the UK and USA. Nat Hum Behav. 2021 Mar;5(3):337-348. doi: 10.1038/s41562-021-01056-1. Epub 2021 Feb 5. PMID 33547453
- [Background] MacDonald NE; SAGE Working Group on Vaccine Hesitancy. Vaccine hesitancy: Definition, scope and determinants. Vaccine. 2015 Aug 14;33(34):4161-4. doi: 10.1016/j.vaccine.2015.04.036. Epub 2015 Apr 17. PMID 25896383